CLINICAL TRIAL: NCT04255914
Title: "Clinical Evaluation of Root Coverage in Miller Class III Gingival Labial Recessions Treated With Interdisciplinary Periodontic - Orthodontic Therapy: A Randomized Controlled Clinical Trial"
Brief Title: Root Coverage in Miller Class III Recessions by Perio-ortho Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sakshi PGIDS/IEC/2019/27
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Orthodontics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root coverage procedure along with orthodontic treatment (Experimental): subepithelial connective tissue graft and orthodontic levelling and alignment
  Interventions: Procedure: Periodontal plastic surgery procedure and orthodontic treatment
- Root coverage procedure only (Active Comparator): sub epithelial connective tissue graft procedure for recession coverage
  Interventions: Procedure: Periodontal plastic surgery procedure

INTERVENTIONS:
Procedure: Periodontal plastic surgery procedure and orthodontic treatment — subepithelial connective tissue graft and orthodontic tooth levelling and alignment
  Arms: Root coverage procedure along with orthodontic treatment
Procedure: Periodontal plastic surgery procedure — subepithelial connective tissue graft procedure
  Arms: Root coverage procedure only

SUMMARY:
To predict root coverage in Miller class III gingival recessions in chronic periodontitis patients using interdisciplinary orthodontic-periodontal surgical treatment as compared to periodontal surgical treatment alone.

DETAILED DESCRIPTION:
INTRODUCTION Gingival recession is defined as the displacement of the gingival margin apical to the cementoenamel junction with exposure of the root surface to the oral environment.The resulting root surface exposure often causes aesthetic concerns, dentin hypersensitivity and increased susceptibility to root caries.

In 1985, Miller proposed a classification of gingival recession and according to Miller, root coverage is more predictable and more successful with class I and class II defects (upto 100%). However, only partial coverage can be obtained with Miller class III (50-70%) and no coverage can be done in class IV defects (0-10%). Miller class III recession is defined as marginal tissue recession which extends to or beyond the mucogingival junction. There is bone or soft tissue loss interdentally or malpositioning of the tooth.

The two primary etiological factors in the pathogenesis of gingival recession are periodontal diseases and mechanical trauma. Other predisposing factors associated with this condition are labial orthodontic tooth movement, bone dehiscence and fenestration, thin gingival biotype and malpositioning of the teeth.Among the numerous orthodontic treatment procedures and modalities, the proclination of incisors outside their dentoalveolar envelop has been considered as a source of gingival recession for years. It has been assumed that presence of bony dehiscence before the beginning of orthodontic therapy is a prerequisite for the development of gingival recession.However, there are very few clinical studies that have actually investigated the relationship between orthodontic tooth movement and gingival recession. Some of them have shown gingival recession to be associated with proclination of mandibular incisors, whereas others have found no such correlation.

Successful coverage of exposed roots for aesthetic and functional reasons has been the objective of various mucogingival surgeries. Pedicle soft tissue grafts (double-papillae, coronally and laterally positioned flaps), free gingival grafts, subepithelial connective tissue grafts, guided tissue regeneration and acellular dermal matrix allografts combined with coronally positioned flaps are the main surgical techniques that have been used to obtained the root coverage. Certain orthodontic movements such as bodily movements have been found to be effective at improving gingival recession.However, it is necessary to have a sufficient amount of keratinised gingiva for orthodontic movement to contribute to reduction of gingival recession. According to Wennstrom et al., the width of keratinised tissue influences the outcome of root coverage; thick tissues and large amounts of keratinised tissue have a favourable prognosis.Historically, gingival augmentation was done to recreate the zone of attached gingiva. Many still believe that attached gingiva is more suitable to withstand the trauma of mastication and tooth brushing. Huang et al. concluded that the initial gingival thickness is the most decisive factor regarding the accomplishment of complete root coverage.Management of gingival recession in orthodontic patients remains unclear, since no higher level of evidence is available. According to Cortellini et al., there is no information as to whether tooth position (buccal or lingual) might influence the outcome of surgical mucogingival procedures.Esteibar et al. stated that it seems likely that the attainment of complete root coverage in cases traditionally classified as Miller class III and considered less severe would not occur by chance, but rather be a response to some preoperative clinical variables and intraoperative measures.Therefore, an interdisciplinary treatment approach is imperative for some of the challenging and complex dental situations in order to improve aesthetics and prognosis.

Predictable coverage of deep isolated Miller class III anterior gingival recessions is one of the most challenging endeavors in plastic-aesthetic periodontal surgery and limited data is available in the literature. Furthermore, most studies have only evaluated treatment of Miller class I and II isolated mandibular recessions, and limited information is available on the treatment of isolated mandibular Miller class III defects.A thorough search of literature revealed a very modest level of evidence -one study with prospective and retrospective data collection and the other one is a retrospective study. In both of the studies, gingival augmentation surgery was carried out before the orthodontic intervention. It is obvious that a well designed clinical trial needs to be conducted so as to explore this issue. Therefore, the current study has been designed so as to predict how much root coverage could be achieved by interdisciplinary orthodontic and periodontal surgical treatment approach in comparison to periodontal surgical procedure alone in Miller class III gingival recession.

Material and Methods

STUDY DESIGN SETTING :

The present prospective, analytical, randomized controlled clinical trial will be conducted in the Department of Periodontology in collaboration with the Department of Orthodontics, Postgraduate Institute of Dental Sciences, Rohtak.

STUDY PERIOD: February 2020 to April 2021

STUDY SUBJECTS: Systemically healthy individuals having slight crowding in the anterior region, with at least one tooth having gingival recession in the same region.

SAMPLE SIZE: A sample size of total 32 participants was calculated by using basic formula of sample size calculation with an effect size of 1 (0.5 mm of improvement in mean levels of gingival margins with a standard deviation of 0.5 in the selected population), α = 0.05 and power = 0.80. In order to compensate for any possible attrition of participants during the course of the study, a total of 36 participants will be recruited for the present study.

METHOD OF RECRUITMENT:

Participants will be enlisted from the regular outpatient department of the Department of Periodontics and Oral Implantology, Department of Orthodontics and Department of Oral Medicine Diagnosis and Radiology after screening on the basis of inclusion and exclusion criteria and their consent for study treatment plan. All participants will be given an outline of the study design and all patient-specific considerations and concerns will be properly addressed. All participants will be required to provide written informed consent.

RANDOMIZATION:

All patients enrolled in the study will be further randomly divided into the following two groups using the random allocation software system by block randomization of 2X2.

1. Root coverage procedure along with orthodontic treatment (Test group) - scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage will be done using subepithelial connective tissue graft. Orthodontic treatment will be initiated 3 months following the grafting procedure.
2. Root coverage procedure only (Control group) - scaling and root planing will be performed and after resolution of periodontal inflammation, root coverage will be done using sub epithelial connective tissue graft.

INTERVENTION:

SCALING AND ROOT PLANING: Full mouth scaling and root planing will be performed using ultrasonic instruments and hand instruments as needed.

PERIODONTAL SURGICAL PROCEDURE:

After administration of local anaesthesia, recipient bed will be prepared in the recession region and connective tissue graft will be procured from the palate or tuberosity area for root coverage procedure. The palatal wound will be sutured to obtain primary wound closure. The connective tissue graft will then be placed on the denuded root surface and sutured to the periosteum using resorbable sutures. This will be followed by periodontal dressing placement.

POST-OPERATIVE CARE:

* Suitable antibiotics and analgesics will be prescribed for 5 days.
* Instructions will be given for gentle brushing with a soft toothbrush and reinstructed for proper oral hygiene maintenance.

The dressing and sutures will be removed after 7-10 days. The patient will be recalled for examination weekly for upto 1 month after surgery and again at 3 months, 6 months and 9 months or till the end of levelling and alignment in test group.

ORTHODONTIC PROCEDURE: All the patients will be treated with the same fixed mechanotherapy. Alignment and levelling will be done using MBT 0.022 slot with wire sequencing as follow: 0.014 NiTi, 0.016 NiTi, 0.018 NiTi,0.018 SS, 0.017*0.025 SS. Biomechanics will include the application of light continuous and well-balanced forces. Oral hygiene motivation and maintenance will be done during the entire course of orthodontic treatment. Once the levelling and alignment (approximately 6-8 months) of teeth has been completed, parameters will be recorded for both test group and control group.

FOLLOW UP: After enrollment, participants will be instructed about oral hygiene maintenance and undergo nonsurgical periodontal treatment in the form of scaling and root planing. All baseline parameters will be recorded 4-6 weeks after SRP (once gingival inflammation is resolved). Placement of subepithelial connective tissue graft will be done in the Test group and participants will be recalled after 3 months for recording all parameters. This will be followed by initiation of orthodontic treatment. Among the Control group participants, subepithelial connective tissue graft will be placed after resolution of gingival inflammation (4-6 weeks after SRP). Both groups will be re-evaluated and undergo recording of all parameters at the end of final treatment.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA:

* Age 18-35 years.
* Anterior tooth displaying Miller's class III gingival recession / RT2, with malposition which required orthodontic treatment.
* Presence of clinically identifiable cementoenamel junction.
* Patient demonstrating compliance for maintaining good oral hygiene after Phase I treatment (evaluated using plaque index < 1%).

Exclusion Criteria:

* EXCLUSION CRITERIA:

  * Patient having any systemic illness (such as diabetes, hyperthyroidism, autoimmune diseases, etc.) that is known to affect the periodontium or outcome of periodontal treatment.
  * Aggressive Periodontitis.
  * Patients taking medications which are known to interfere with periodontal wound healing such as corticosteroids, calcium channel blockers or long-term NSAIDS.
  * Pregnant or lactating women.
  * Cervically restored teeth and the presence of severe cervical abrasion, erosion or root caries.
  * Non vital tooth.
  * Current and past smokers.
  * Patients with oral piercing.
  * Mobile teeth.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
root coverage | 12 months
  percentage of root coverage by calculating recession depth preoperatively and postoperatively

SECONDARY OUTCOMES:
bleeding on probing | 12 months
  evaluating bop preoperative and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: SAKSHI MALHOTRA, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES,ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

REFERENCES:
- [Derived] Malhotra S, Tewari S, Sharma R, Sharma RK, Tanwar N, Arora R. Clinical evaluation of root coverage in Miller class III/RT2 labial gingival recession treated with interdisciplinary periodontal-orthodontic therapy: a randomized controlled clinical trial. J Periodontal Implant Sci. 2024 Aug;54(4):265-279. doi: 10.5051/jpis.2204100205. Epub 2023 Nov 20. PMID 38290996